CLINICAL TRIAL: NCT02004496
Title: Randomized Controlled Single-blind Trial to Evaluate the Mobile Tracking of Symptoms in Ambulatory Breast Cancer Patients
Acronym: PatAPP1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Termination due to relevant update of the operation system. Adaption of the application was not foreseen in the intervention study.
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PatAPP1, Version 1.3
Record Dates: First submitted 2013-11-25; First posted 2013-12-09 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A: no app (No Intervention): no use of an mobile application while treatment
- Group B: only app (Active Comparator): Patients, who use independently the mobile application named Consilium without involvement of the physician.
  Interventions: Device: Consilium
- Group C: app and physician (Active Comparator): Patients use the mobile application named Consilium in collaboration with the physician.
  Interventions: Device: Consilium

INTERVENTIONS:
Device: Consilium — Patients use a mobile application to track their subjective well-being and adverse events (AE) while ambulant chemotherapy. The mobile app supports the patients in the structured and standardized entry of their data and is developed specifically for this study.
  Other Names: mobile application
  Arms: Group B: only app; Group C: app and physician

SUMMARY:
Health care has an increasingly demand for mobile applications (App), but studies are rare, which explore the added value and benefits for patient and physician. Patients in different disease groups or physicians from different specialties are likely to have different demands. Research should focus on selected groups to better understand their individual demands. Our study intends to identify the added value of mobile symptom tracking in a selected subgroup of patients. We designed an App for breast cancer patients, who receive ambulant chemotherapy in a breast center. The patients track regularly their well-being and adverse events (AE) with the smartphone- or web-app and share it with the physician in the medical consultation. The data entry was designed to meet patient needs based on previous usability testing.

The reporting of AE and well-being are standardized according to the definitions by CTCAE 4.0 and ECOG-Index to ensure the reliability of patient self-reporting.

The primary outcomes are the number of reported AE, the influence on their subjective well-being and the acceptance of context specific information. We will include 150 participants in this study. The calculated power is 91% respectively 80% for a 10 % improvement of well-being and a 2.2 increase of detected AEs.

The results will be compared to patients without App and to patients with App but without shared information.

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* female
* 18 years old and older
* German speaking
* written informed consent
* beginning of intravenous chemotherapy in the breast care center
* diagnosis breast cancer
* personal smartphone (own device)

Exclusion criteria:

- patients who did not meet the inclusion criteria or if compliance could be questioned, e.g. due to a psychiatric illness or personal life.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-12; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of reported Adverse Events | 5-6 weeks for each patient
  Patients report their adverse events independently in a mobile app for a period of 3 cycles of chemotherapy. The reporting of AE and well-being are standardized according to the definitions by CTCAE 4.0 and ECOG-Index to ensure the reliability of patient self-reporting. Medical consultations take place periodically every 2-3 weeks. Planned medical consultations: start-consultation with the begin of chemotherapy, first consultation before the 2nd chemotherapy cycle and second (final) consultation before the 3rd chemotherapy cycle.
  The observation time of each patient is 5-6 weeks.
influence on patients subjective well-being | 5-6 weeks for each patient
  Patients report their adverse events independently in a mobile app for a period of 3 cycles of chemotherapy. The reporting of AE and well-being are standardized according to the definitions by CTCAE 4.0 and ECOG-Index to ensure the reliability of patient self-reporting. Medical consultations take place periodically every 2-3 weeks. Planned medical consultations: start-consultation with the begin of chemotherapy, first consultation before the 2nd chemotherapy cycle and second (final) consultation before the 3rd chemotherapy cycle.
  The observation time of each patient is 5-6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Trojan, MD, Principal Investigator — University Hospital Zurich, Clinical Pharmacology and Toxicology
Locations (1):
- University Hospital Zurich, Clinical Pharmacology and Toxicology, Zurich, Switzerland

REFERENCES:
- [Derived] Trojan A, Roth S, Atassi Z, Kiessling M, Zenhaeusern R, Kadvany Y, Schumacher J, Kullak-Ublick GA, Aapro M, Eniu A. Comparison of the Real-World Reporting of Symptoms and Well-Being for the HER2-Directed Trastuzumab Biosimilar Ogivri With Registry Data for Herceptin in the Treatment of Breast Cancer: Prospective Observational Study (OGIPRO) of Electronic Patient-Reported Outcomes. JMIR Cancer. 2024 Apr 4;10:e54178. doi: 10.2196/54178. PMID 38573759
- [Derived] Trojan A, Battig B, Mannhart M, Seifert B, Brauchbar MN, Egbring M. Effect of Collaborative Review of Electronic Patient-Reported Outcomes for Shared Reporting in Breast Cancer Patients: Descriptive Comparative Study. JMIR Cancer. 2021 Mar 17;7(1):e26950. doi: 10.2196/26950. PMID 33729162
- [Derived] Egbring M, Far E, Roos M, Dietrich M, Brauchbar M, Kullak-Ublick GA, Trojan A. A Mobile App to Stabilize Daily Functional Activity of Breast Cancer Patients in Collaboration With the Physician: A Randomized Controlled Clinical Trial. J Med Internet Res. 2016 Sep 6;18(9):e238. doi: 10.2196/jmir.6414. PMID 27601354